CLINICAL TRIAL: NCT00053846
Title: Buspirone in Reducing Shortness of Breath in Patients With Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Gary Morrow, Director, URCC CCOP Research Base, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000269487; U10CA037420 (NIH); URCC U1701 (Other: University of Rochester)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Dyspnea; Pulmonary Complications; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: dyspnea; pulmonary complications; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Dyspnea | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- buspirone hydrochloride (Experimental): buspirone hydrochloride
  Interventions: Drug: buspirone hydrochloride
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: buspirone hydrochloride — The dose of buspirone will be 10 mg taken by mouth at bedtime for 3 days, then twice each day, in the morning and at bedtime for the remainder of the 28 day study period
  Arms: buspirone hydrochloride
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
RATIONALE: Buspirone may be effective in reducing dyspnea (shortness of breath) in patients with cancer who are undergoing chemotherapy.

PURPOSE: Randomized clinical trial to study the effectiveness of buspirone in reducing shortness of breath in patients who are undergoing chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the degree to which buspirone can decrease the sensation of dyspnea in patients with malignant disease.
* Estimate the incidence of dyspnea in patients seen in community oncology practice settings.
* Investigate interrelationships of fatigue, depression, anxiety, and patient report of dyspnea.
* Assess the quality of life of patients treated with this drug.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center (CCOP site). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning on day 7 of chemotherapy, patients receive oral buspirone once a day for 3 days and then twice daily for up to 28 days.
* Arm II: Patients receive oral placebo as in arm I. Dyspnea is assessed at baseline. Dyspnea, mood, fatigue, depression, anxiety, and quality of life are assessed within 5-7 days before chemotherapy and immediately following therapy.

PROJECTED ACCRUAL: A total of 376 patients (188 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Treatment includes the following scenarios:

  * May have had prior chemotherapy course(s)
  * Scheduled to receive at least 2 courses of chemotherapy

    * Courses may include multiple treatment days such as days 1-5 or day 1-day 8 regimens and may include oral regimens
* Dyspnea as a symptom within the past 5 days (defined by a score of at least grade 2 on the Modified Medical Research Council Dyspnea Scale)

  * All underlying causes of dyspnea have received medical treatment per best clinical judgement of treating physician

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Eastern Cooperative Oncology Group 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Adequate hepatic function (determined by treating oncologist)

Renal

* Adequate renal function (determined by treating oncologist)

Cardiovascular

* Adequate cardiac function (determined by treating oncologist)

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No history of mania or seizures
* No prior hospitalization for any psychiatric condition
* No prior hypersensitivity to buspirone
* Able to swallow medication

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Concurrent radiotherapy allowed

Surgery

* Not specified

Other

* At least 2 weeks since prior and no concurrent monoamine oxidase inhibitors (MAOIs)
* Concurrent narcotic medications allowed
* Concurrent benzodiazepine medications allowed
* Concurrent serotonin reuptake inhibitors allowed
* No concurrent alcohol

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2002-11; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bushunow, MD, Study Chair — University of Rochester
Locations (15):
- United States (15):
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Northwest, Tacoma, Washington
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Treatment with placebo will be one tablet taken by mouth at bedtime for 3 days, then twice each day, in the morning and at bedtime for the remainder of the study period.
Period: Overall Study
Arm/Group | Buspirone Hydrochloride | Placebo
Started | 213 | 219
Completed | 187 | 192
Not Completed | 26 | 27
Not completed — Changed mind | 8 | 13
Not completed — Became too ill | 8 | 7
Not completed — Expired | 5 | 0
Not completed — Became ineligible | 3 | 1
Not completed — Did not return data | 1 | 2
Not completed — Quit due to side effects | 1 | 3
Not completed — Pills too large | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buspirone Hydrochloride | Placebo | Total
Number analyzed (Participants) | 187 | 192 | 379
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (10.3) | 64.0 (9.4) | 63.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 95 | 195
  Male | 87 | 97 | 184
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 181 | 189 | 370
  Unknown or Not Reported | 6 | 1 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  White | 166 | 171 | 337
  African American | 19 | 20 | 39
  Other | 2 | 1 | 3
Marital Status [Number; unit: participants]
  Married | 127 | 126 | 253
  Not Married | 60 | 66 | 126
Education [Number; unit: participants]
  Beyond High School | 76 | 78 | 154
  High School or Less | 111 | 114 | 225
History of chronic obstructive pulmonary disease (COPD) [Number; unit: participants]
  Yes | 28 | 69 | 97
  No | 159 | 123 | 282
Tumor Site [Number; unit: participants]
  Lung | 114 | 118 | 232
  Breast | 25 | 27 | 52
  Gastrointestinal | 18 | 17 | 35
  Other | 30 | 30 | 60
Tumor Stage [Number; unit: participants]
  I | 10 | 12 | 22
  II | 17 | 18 | 35
  III | 49 | 53 | 102
  IV | 103 | 102 | 205
  Unknown | 8 | 7 | 15
O2 Cost Diagram (OCD) [Mean (Standard Deviation); unit: units on a scale] — Oxygen Cost Diagram (OCD) is used to evaluate dyspnea on exertion and activities of daily living. OCD is a visual analog scale for quantifying a patient's evaluation of tolerance for exertion. It corresponds to the oxygen requirements at different activity levels. It is presented as a score ranging from 2 (i.e.; even sleeping induces exertion) to 14 (i.e., unable to walk briskly uphill). Higher scores indicate fewer limitations due to dyspnea.
  units on a scale | 8.70 (2.6) | 8.43 (2.6) | 8.56 (2.6)
Modified Medical Research Council Dyspnea Scale (MMRCDS) Grade [Number; unit: participants] — The Modified Medical Research Council Dyspnea Scale (MMRCDS) Grade is assessed on a 5-point scale with a range of 0 to 4. Grade 0 (I only get breathless with strenuous exercise) to Grade 4 (I am too breathless to leave the house or I am breathless when dressing). Higher scores are less favorable.
  participants
    0 | 4 | 2 | 6
    1 | 21 | 23 | 44
    2 | 77 | 80 | 157
    3 | 61 | 54 | 115
    4 | 22 | 32 | 54
    Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Dyspnea as Measured by Oxygen Cost Diagram (OCD)
Description: OCD was used to evaluate dyspnea on exertion and activities of daily living. OCD is a visual analog scale for quantifying a patient's evaluation of tolerance of exertion, which corresponds to oxygen requirements at different activity levels. It is measured as a score of 2 (sleeping) to 14 (brisk walking uphill). HIgher scores indicate fewer limitations due to dyspnea.
Time Frame: 28 days after beginning study drug or placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone Hydrochloride | Placebo
Number analyzed (Participants) | 187 | 192
units on a scale | 8.98 (2.85) | 9.32 (2.62)
Statistical Analysis 1: Comparison: Buspirone Hydrochloride vs Placebo; H0: The true difference in means is equal to zero. Ha: The true difference in means is not equal to zero; Test type: Superiority or Other; p = 0.080, ANCOVA; Mean Difference (Final Values) = -0.483, 95% CI 2-sided [-1.020 to 0.0576], Standard Error of Mean 0.2750 — Multiple Imputation (MI) used for estimates. MICE software in R was used to generate 100 imputed datasets. ANCOVA was run on each, and results were pooled

ADVERSE EVENTS:
Arm/Group | Buspirone Hydrochloride | Placebo
Serious Adverse Events (participants affected / at risk) | 3/213 | 3/219
Other Adverse Events (participants affected / at risk) | 13/213 | 10/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buspirone Hydrochloride (N=213) | Placebo (N=219)
Esophagitis (Gastrointestinal disorders) | 0 | 1
Breathlessness & Chest Pressure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anemia & pleural effusion, inc SOB (General disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Scrotal pain/swelling; hypoxia; death (General disorders) | 0 | 1
Death (General disorders) | 2 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buspirone Hydrochloride (N=213) | Placebo (N=219)
Dizziness, confusion; insomnia (Nervous system disorders) | 2 | 2
GI Bleed (Gastrointestinal disorders) | 0 | 1
Aching hands and back (General disorders) | 0 | 1
Nausea and vomitting (Gastrointestinal disorders) | 3 | 1
Disease progression (General disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 3
Confusion (Nervous system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Shakes and tremors (General disorders) | 0 | 2
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pneumonia/bronchitis (Infections and infestations) | 1 | 0
Low platelet count (Blood and lymphatic system disorders) | 1 | 0
Hypoxemia (Blood and lymphatic system disorders) | 1 | 0
Orthostatis hypotension (Blood and lymphatic system disorders) | 0 | 1
Thrombosis (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No